CLINICAL TRIAL: NCT05422157
Title: Evaluation of the Inter-center Variability of the Measurement of Thrombin Generation by the ST Genesia System
Acronym: EVIGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LEBRETON 3 (EVIGE); 2021-A01971-40 (Other: 2021-A01971-40)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Patients Without a Medical History of Thrombosis or Hemorrhage; Hemophilic Patient; Patient With FV Leiden Mutation; Patient With Cirrhosis; Patient on Anticoagulant
Keywords: Coagulation; Variability; Hemostasis; Thrombin generation
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: No intervention. Collection of additional blood volume (50 mL) during blood tests provided as part of the usual medical care.
- Hemophilia: No intervention. Collection of additional blood volume (50 mL) during blood tests provided as part of the usual medical care.
- FV Leiden: No intervention. Collection of additional blood volume (50 mL) during blood tests provided as part of the usual medical care.
- Cirrhosis: No intervention. Collection of additional blood volume (50 mL) during blood tests provided as part of the usual medical care.
- Anticoagulation: No intervention. Collection of additional blood volume (50 mL) during blood tests provided as part of the usual medical care.

SUMMARY:
The thrombin generation test is a global test for the study of coagulation that allows the fine study of the balance between procoagulant and anticoagulant factors. For many years, it has been performed in laboratories by semi-automated techniques, sometimes using in-house reagents, which led to a high variability and did not allow multicenter studies. Recently, an automated device for the evaluation of thrombin generation has been placed on the market (ST-Genesia), allowing a better standardization of the technique. In order to allow multicenter studies, which are essential for the routine positioning of the thrombin generation test, the inter-center variability must be evaluated, as a priority, in the pathologies for which the test is routinely positioned.

Thrombin generation (TG) assays are long-established research tools in hemostasis. They are used for both fundamental and clinical research, but a multiplicity of test methodologies limits the large adoption of TG due to the variability of results despite the attempts to standardize practices.

Several publications already exist to evaluate its analytical performances, and thereby demonstrate that the test automation also allows its democratization to reach acceptable performances It also enables the evaluation of the device in various indications such as, for example, the evaluation of the effect of direct oral anticoagulants or the evaluation of the risk of breast cancer recurrence.

The confirmation of these anterior results allows further clinical investigations in larger cohorts. However, the absence of interchangeability between the two systems indicates that the results will need to be more rugged through multicenter studies on ST Genesia.

DETAILED DESCRIPTION:
A preliminary step in the development of multi-center protocols is to confirm that inter-center variability is acceptable on ST Genesia, and even more acceptable than it was on Calibrated Automated Thrombogram (CAT). Since the variability of the results can be attributed to analytical, pre-analytical and inter-individual biological variabilities, it has been agreed that the evaluation that we will conduct will focus only on the analytical variability and will therefore be carried out on the same samples, collected and prepared in the sponsoring center of the study, and distributed in the form of frozen aliquots to the different co-investigating centers.

The evaluation of this inter-center variability of this new device will allow, if satisfactory, to propose multicenter studies. These are essential in order to position the thrombin generation test in routine in these various promising clinical contexts.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, male or female
* Affiliated to a social security system
* In capacity to express informed consent to participate in research
* Control group: 5 men, 5 women without oral contraception, 5 women with oral contraception and apparently healthy with a respect to hemostasis (no history of thrombosis or significant bleeding on examination)
* Hemophilia groups: - 5 hemophiliacs A (treated or untreated), with predictable FVIII:C levels between < 1% and 40%.
* 5 hemophiliacs B (treated or not), with predictable FIX:C levels between < 1% and 40%.
* FV Leiden group: 5 patients known to be heterozygous or homozygous for the R506Q mutation of the F5 gene (the so-called "Factor V Leiden" mutation)
* Cirrhosis group: - 5 patients with Child-Pugh A
* 5 patients with Child-Pugh B
* 5 patients with Child-Pugh C
* Anticoagulation group: - 5 patients on anti-vitamin K therapy for at least 1 month, with INR between 2 and 4
* 5 patients on apixaban for at least 1 week
* 5 patients on rivaroxaban for at least 1 week
* 5 patients on dabigatran for at least 1 week
* 5 patients on low molecular weight heparin for at least 1 day

Exclusion Criteria:

* Refusal to participate
* Patient under protective measures (guardianship, curatorship) or under judicial protection
* Minor patients
* Moderate to end-stage renal failure
* Proven inflammatory state/infectious syndrome (body temperature > 38°C and/or clinical signs suggestive of infection) during or in the week prior to collection, at the discretion of the investigator
* Transfusion in the week prior to collection
* Pregnant or breastfeeding woman
* Contraception by estrogen-progestin, except for the control group concerned
* Anticoagulation of less than one week, except for the anticoagulation group
* Control group: - Presence of drug treatment known to interfere with hemostasis
* Presence of a pathology known to interfere with hemostasis such as renal or hepatic insufficiency
* Presence of a history of venous thromboembolic disease or diagnosed hemorrhagic disease
* Predicted inclusion hemoglobin level < 7g/L
* Hemophilic groups: - Presence of anti FVIII or anti FIX inhibitors
* Treatment with emicizumab
* Predicted inclusion hemoglobin level < 7g/L
* FV Leiden group: - Presence of anticoagulant therapy at the time of collection
* Predicted baseline hemoglobin < 7g/L
* Anticoagulation group: - Anticoagulant therapy not stabilized as determined by the practitioner
* Presence of a therapeutic relaunch in progress
* Hemoglobin at predicted inclusion < 9-10g/L
* Cirrhosis group: Predicted inclusion hemoglobin level < 7g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient taken care of at the Clermont-Ferrand University Hospital
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the inter-center analytical variability of the thrombin generation measurement on ST Genesia, on different types of normo-, hypo- or hyper-coagulable samples. | at the time of inclusion
  Assessing the analytical variability of the thrombin generation measurement on ST Genesia, compared to that observed on CAT, on different groups of patients

SECONDARY OUTCOMES:
Assessment of inter-center analytical variability on ST Genesia related to different reagent lots, for centers with multiple reagent lots. | at the time of inclusion
  Measure of the thrombin generation in absolute value
Comparing the analytical variability between centers observed on the same samples on the reference system, the Calibrated Automated Thrombogram, for centers also equipped with this device | at the time of inclusion
  Investigate the differences between thrombin generation measurements on CAT and ST genesia

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Lebreton, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Hemker HC. Recollections on thrombin generation. J Thromb Haemost. 2008 Feb;6(2):219-26. doi: 10.1111/j.1538-7836.2008.02864.x. Epub 2007 Dec 10. PMID 18088345
- [Background] Baglin T. The measurement and application of thrombin generation. Br J Haematol. 2005 Sep;130(5):653-61. doi: 10.1111/j.1365-2141.2005.05612.x. PMID 16115120
- [Background] de Laat-Kremers RMW, Ninivaggi M, Devreese KMJ, de Laat B. Towards standardization of thrombin generation assays: Inventory of thrombin generation methods based on results of an International Society of Thrombosis and Haemostasis Scientific Standardization Committee survey. J Thromb Haemost. 2020 Aug;18(8):1893-1899. doi: 10.1111/jth.14863. Epub 2020 Jun 3. PMID 32319140
- [Background] Dargaud Y, Wolberg AS, Luddington R, Regnault V, Spronk H, Baglin T, Lecompte T, Ten Cate H, Negrier C. Evaluation of a standardized protocol for thrombin generation measurement using the calibrated automated thrombogram: an international multicentre study. Thromb Res. 2012 Dec;130(6):929-34. doi: 10.1016/j.thromres.2012.07.017. Epub 2012 Aug 19. PMID 22909826
- [Background] Perrin J, Depasse F, Lecompte T; French-speaking CAT group and under the aegis of GEHT; French-speaking CAT group (all in France unless otherwise stated):; French-speaking CAT group all in France unless otherwise stated. Large external quality assessment survey on thrombin generation with CAT: further evidence for the usefulness of normalisation with an external reference plasma. Thromb Res. 2015 Jul;136(1):125-30. doi: 10.1016/j.thromres.2014.12.015. Epub 2014 Dec 24. PMID 25563679
- [Background] Calzavarini S, Brodard J, Quarroz C, Maire L, Nutzi R, Jankovic J, Rotondo LC, Giabbani E, Fiedler GM, Nagler M, Angelillo-Scherrer A. Thrombin generation measurement using the ST Genesia Thrombin Generation System in a cohort of healthy adults: Normal values and variability. Res Pract Thromb Haemost. 2019 Jul 18;3(4):758-768. doi: 10.1002/rth2.12238. eCollection 2019 Oct. PMID 31624796
- [Background] Douxfils J, Morimont L, Bouvy C, de Saint-Hubert M, Devalet B, Devroye C, Dincq AS, Dogne JM, Guldenpfennig M, Baudar J, Larock AS, Lessire S, Mullier F. Assessment of the analytical performances and sample stability on ST Genesia system using the STG-DrugScreen application. J Thromb Haemost. 2019 Aug;17(8):1273-1287. doi: 10.1111/jth.14470. Epub 2019 May 31. PMID 31063645
- [Background] Foulon-Pinto G, Jourdi G, Perrin J, Abdoul J, Paris G, Gouin-Thibault I, Curis E, Lecompte T, Siguret V. Study of thrombin generation with St Genesia to evaluate xaban pharmacodynamics: Analytical performances over 18 months. Int J Lab Hematol. 2021 Aug;43(4):821-830. doi: 10.1111/ijlh.13443. Epub 2020 Dec 28. PMID 33369212
- [Background] Mori F, Genuardo C, Nannizzi S, Farina C. Intra- and interassay variations of two thrombin generation methods. Int J Lab Hematol. 2021 Aug;43(4):O218-O220. doi: 10.1111/ijlh.13524. Epub 2021 Mar 24. No abstract available. PMID 33759358
- [Background] Metze M, Pfrepper C, Kloter T, Stobe S, Siegemund R, Siegemund T, Edel E, Laufs U, Petros S. Inhibition of thrombin generation 12 hours after intake of direct oral anticoagulants. Res Pract Thromb Haemost. 2020 Apr 23;4(4):610-618. doi: 10.1002/rth2.12332. eCollection 2020 May. PMID 32548560
- [Background] Gomez-Rosas P, Pesenti M, Verzeroli C, Giaccherini C, Russo L, Sarmiento R, Masci G, Celio L, Minelli M, Gamba S, Tartari CJ, Tondini C, Giuliani F, Petrelli F, D'Alessio A, Gasparini G, Labianca R, Santoro A, De Braud F, Marchetti M, Falanga A; HYPERCAN Investigators. Validation of the Role of Thrombin Generation Potential by a Fully Automated System in the Identification of Breast Cancer Patients at High Risk of Disease Recurrence. TH Open. 2021 Feb 10;5(1):e56-e65. doi: 10.1055/s-0040-1722609. eCollection 2021 Jan. PMID 33585786
- [Background] Talon L, Sinegre T, Lecompte T, Pereira B, Massoulie S, Abergel A, Lebreton A. Hypercoagulability (thrombin generation) in patients with cirrhosis is detected with ST-Genesia. J Thromb Haemost. 2020 Sep;18(9):2177-2190. doi: 10.1111/jth.14963. Epub 2020 Jul 23. PMID 32558351